CLINICAL TRIAL: NCT05612594
Title: Adipose Dysfunction, Imaging, Physiology, and Outcomes With SGLT2i's for Sleep Apnea: The ADIPOSA Study
Brief Title: Adipose Dysfunction, Imaging, Physiology, and Outcomes With Sodium Glucose Cotransporter 2 Inhibitor (SGLT2i) for Sleep Apnea: The ADIPOSA Study
Acronym: ADIPOSA
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Case Western Reserve University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2000033371
Record Dates: First submitted 2022-11-03; First posted 2022-11-10 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Sleep Apnea
MeSH Terms: conditions — Sleep Apnea Syndromes | interventions — bexagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, study personnel, and outcomes adjudicators will be blinded to the treatment assignment until the end of study procedures and database lock. Blinding codes will be broken at the end of the trial. Blinding codes will only be broken before the end of trial if a participant develops a serious adverse event requiring knowledge of the treatment allocation. At such time, the participant will be considered to have completed the trial and will not undergo any further trial treatment but may be asked to undergo assessment of trial endpoints when feasible. Whenever a code is broken, the person breaking the code must complete the unblinding form in Redcap. If the participant should be withdrawn following a code break, a withdrawal session should be completed in the computerized randomization system.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bexagliflozin (Experimental): Bexagliflozin once daily for 6 months
  Interventions: Drug: Bexagliflozin 20 mg
- Placebo (Placebo Comparator): Placebo once daily for 6 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bexagliflozin 20 mg — 15mg once daily
  Arms: Bexagliflozin
Drug: Placebo — matching placebo once daily
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to test if bexagliflozin lowers the sleep apnea severity in adults who are overweight or obese with moderate to severe obstructive sleep apnea (OSA) compared with a placebo (look-alike substance that contains no active drug).

The main question it aims to answer is:

* If SGLT2i will reduce anatomic and physiologic traits, clinical measures of OSA and sleep deficiency in participants
* If improvement in clinical measures are because of improvement in the anatomic and physiologic traits.

Participants will be placed on either drug or placebo and get routine normal care for 6 months. At the start and end of the study, participants will undergo different clinical measurements to see if the drug makes the sleep apnea better.

DETAILED DESCRIPTION:
The primary objective of this study is to determine whether bexagliflozin 20 mg once daily compared with placebo reduces the apnea hypopnea index (AHI) in adults with overweight or obesity with moderate to severe OSA.

The secondary objectives of this study are to determine whether bexagliflozin 20 mg once daily compared with placebo (a look-alike substance that contains no active drug):

* reduces visceral and neck fat and upper airway soft tissue structure volumes and increases airway caliber
* reduces Critical closing pressure
* reduces rostral to caudal fluid shifts (measured by neck circumference)
* improves clinical measures of OSA severity and sleep deficiency

This is a 2-center clinical trial of overweight or obese adults (BMI 25-40 kg/m2) diagnosed with moderate to severe OSA, recruited from University Hospitals Cleveland Medical Center (UH) and Yale New Haven Health (YNHH). Participants will be randomized to bexagliflozin 20 mg once daily or matching placebo in addition to standard routine clinical care for both groups for 6 months. At baseline and at study end, participants will undergo measurements of anatomic traits using MRI imaging, critical closing pressure, blood-based biomarkers of dysfunctional adiposity, non-anatomic physiologic trait polysomnographic phenotyping, morning neck circumference, clinical measures of sleep apnea severity (apnea hypopnea index (AHI), oxygen desaturation index (ODI), % time with O2sat < 90% (T90)), sleep arousal index (AI)), and measures of sleep deficiency, to evaluate the effects of SGLT2i on the measured phenotypes.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent and stated willingness to comply with all study procedures and availability for the duration of the study
* Overweight or obese (body mass index 25-40 kg/m2)
* Clinically confirmed diagnosis of obstructive sleep apnea by one of the following methods:

  a. Polysomnography: AHI ≥15/hour sleep or b. Home sleep apnea testing: Respiratory event index (REI) ≥15/hour sleep
* AHI: apnea-hypopnea index (apneas + hypopneas / total sleep time in hours)

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Known non-OSA related conditions associated with sleep disordered breathing (e.g., central disorder of hypersomnolence, neurological, neuromuscular, or pulmonary disorder)
* Use of sleep-inducing medications (e.g. benzodiazepines, opiates, barbiturates)
* Type 1 diabetes mellitus
* History of diabetic ketoacidosis
* Known hypersensitivity reaction to bexagliflozin or any of its constituents or any contraindication to bexagliflozin use
* Severe, recurrent urinary tract or genital mycotic infections
* eGFR<30mL/min/1.73m2 at time of or within 4 weeks of enrollment in the study
* Unable to complete/tolerate magnetic resonance imaging (MRI) due to severe claustrophobia or metallic implants.
* Language barrier, mental incapacity, unwillingness or inability to understand.
* Females of childbearing potential who are pregnant, breast-feeding or intend to become pregnant.
* Currently or planning to take a SGLT2i prior to or during enrollment in the study
* Currently or planning to follow a ketogenic diet pattern ("keto diet) prior to or during enrollment in the study
* Currently or planning to follow an active weight loss program (including but not limited to use of supplements, medications, or surgery) prior to or during enrollment in the study
* Currently or planning to follow an intermittent fasting diet plan prior to or during enrollment in the study
* Currently or planning to take a GLP-1 receptor agonist prior to or during enrollment in the study .
* Existing lower limb ulcer (due to diabetes or any cause)
* Existing severe peripheral arterial disease with intermittent claudication and/or prior lower limb revascularization procedure
* Concomitant administration of UGT inducers
* Severe liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2024-03-27 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Change in Apnea hypopnea index (AHI) measured by full ambulatory polysomnography (aPSG) | Baseline and 6 months
  All participants will undergo a full in-home aPSG with a Nox-A1 system, which collects sleep EEG required to determine the physiologic traits and measures of sleep apnea. This is an unattended sleep monitor. The AHI is the number of apneas or hypopneas recorded during the sleep study per hour of sleep. Higher AHI indicates the severity of sleep apnea.

SECONDARY OUTCOMES:
Change in Neck and body fat and lean volume by MRI | Baseline and 6 months
  Participants will undergo standard measurements including height, weight, waist circumference, hip circumference, and neck circumference by MRI to quantify fat and lean tissue composition in the neck and body. Volumetric imaging datasets of the body will be derived by MRI using validated and readily available protocols with rapid scan time to perform precise measurements of total and regional body composition to quantify fat and lean tissue composition in the neck and body. MRI imaging using a 6-minute dual-echo Dixon Vibe protocol, providing water and fat separated volumetric data set covering neck to knees, and a single-slice multi-echo Dixon acquisition for proton density fat fraction (PDFF) assessment in the liver.
Change in Airway caliber by MRI | Baseline and 6 months
  Volumetric imaging datasets of the body derived by MRI using validated and readily available protocols with rapid scan time to perform precise measurements of total and regional body composition to quantify fat and lean tissue composition in the neck and body, including MRI imaging using a 6-minute dual-echo Dixon Vibe protocol, providing water and fat separated volumetric data set covering neck to knees, and a single-slice multi-echo Dixon acquisition for proton density fat fraction (PDFF) assessment in the liver.
Change in Critical closing pressure (Pcrit)/normal ventilatory drive (Vpass) by aPSG | Baseline and 6 months
  Mathematical modeling to determine the patient's ventilatory drive in response to changes in ventilation induced by upper airway obstruction (i.e., apnea/hypopnea). Pharyngeal collapsibility, calculated as the level of ventilation during sleep at normal or eupneic ventilatory drive (Vpassive) and is a valid proxy for critical closing pressure (Pcrit) and a reflection of the impact of the anatomic traits of sleep apnea.
Change in neck circumference | Baseline and 6 months
  Change in neck circumference measured by tape measure. Measuring the change in the evening to morning neck circumference which is a validated measure of caudal to rostral fluid shift. Higher neck circumference indicates an increase in probability of sleep apnea.
Change in Oxygen desaturation index (ODI) measured by aPSG | Baseline and 6 months
  Percent of time with O2 saturation < 90% (T90) recorded during the aPSG
Change in Sleep arousal index (ArI) measured by aPSG | Baseline and 6 months
  Total arousal index (ArI) was defined as the total number of arousals recorded during the aPSG per hour of sleep.
Change in Insomnia Severity Index (ISI) | Baseline, 3 months and 6 months
  The Insomnia Severity Index has seven questions. The seven answers are added up to get a total score. Total scores scale:
  0-7 = No clinically significant insomnia 8-14 = Subthreshold insomnia 15-21 = Clinical insomnia (moderate severity) 22-28 = Clinical insomnia (severe)
Change in Sleep Quality measured by Pittsburgh Sleep Quality Index Form | Baseline, 3 months and 6 months
  This questionnaire contains 19 self-rated questions that are combined to form seven "component" scores, each of which has a range of 0-3 points. In all cases, a score of 0 indicates no difficulty in that area, while a score of 3 indicates severe difficulty. The seven component scores are then added to yield one global score, with a range of 0-21 points, with 0 indicating no difficulty and 21 indicating severe difficulties in all areas.
  The seven component domains are: 1. Subjective sleep quality, 2. Sleep latency, 3. Sleep duration, 4. Habitual sleep efficiency, 5. Step disturbances, 6. Use of sleeping medication, and 7. Daytime dysfunction.
Change in Reduced Morningness Eveningness Questionnaire (MEQ) | Baseline, 3 months and 6 months
  The 5 questions reduced MEQ is a self-assessment questionnaire. Responses to the questions are combined to form a composite score that indicates the degree to which the respondent favors morning versus evening. In Total Score (0-25) higher scores indicate morningness, lower scores indicate eveningness.
Change in Regulatory Satisfaction Alertness Timing Efficiency Duration (RU-SATED) | Baseline, 3 months and 6 months
  Regulatory Satisfaction Alertness Timing Efficiency Duration (RU-SATED) questionnaire. This is a multidimensional metric for sleep health with 6 questions. RU-SATED stands for: regularity of sleep, satisfaction with sleep, alertness during the day, timing of sleep, efficiency of sleep, and duration of sleep. Each question is scored 0, 1, or 2 based on rarely/never, sometimes, usually always responses. The scores are summed, and a higher score indicates better sleep health.
Change in Sleep Deprivation Questionnaire (SDQ) | Baseline, 3 months and 6 months
  The questionnaire is divided into two sections. The first section assesses sleep duration in hours as a weighted average of work night hours and weekend night hours. Sleep deprivation is determined from the reported hours of sleep as follows: ≥7 hours = no sleep deprivation; <7 but ≥5 hours = mild to moderate sleep deprivation; <5 hours = severe sleep deprivation. The second section assesses the circadian timing of sleep by asking questions related to circadian-sleep mismatch; a higher score indicates worse circadian sleep timing.
Change in STOP - Bang questionnaire | Baseline, 3 months and 6 months
  The snoring, tiredness, observed apnea, high BP, BMI, age, neck circumference, and gender (STOP-Bang) questionnaire. The Total Sore 0-8 with higher scores indicating higher risks for obstructive sleep apnea. Affirmative answers get a "1" and the sum of the eight question scores is stratified into low risk for OSA (0-2), moderate risk (3-4), and high risk (5-8).
Change inThe Sleep Apnea Quality of Life Index (SAQLI). | Baseline, 3 months and 6 months
  This is a disease specific quality of life index for OSA in adults. Categories and domains include daily functioning, social interactions, emotional functioning, and symptoms. The scaling of items ranges from "not at all" to "all the time," a seven point scale.
Change in The Epworth Sleepiness Scale (ESS) | Baseline, 3 months and 6 months
  This is a validated scale to assess perceived hypersomnia. Patients are asked to score on a scale of 0 to 3 the likelihood that they would "doze-off" in different scenarios ranging from passes activities to active situations. The low score is zero in the high score is 24. The score of greater than 10 is considered clinically significant hypersomnia.
Change in height. | Baseline and 6 months
  Height measured in cm.
Change in weight. | Baseline and 6 months
  Weight will be recorded to the nearest 0.1 kg using calibrated scales. Weight will be measured in a fasting state with an empty bladder, without shoes and only wearing light clothing.
Change in body mass index (BMI) | Baseline and 6 months
  Body mass index (BMI) is a value derived from the mass (weight) and height of a person. The BMI is defined as the body mass divided by the square of the body height, and is expressed in units of kg/m2, resulting from mass in kilograms and height in metres.
Change in Waist circumference | Baseline and 6 months
  Waist circumference measured in cm.
Change in hip circumference | Baseline and 6 months
  Hip circumference measured in cm.
Change in sleep walking periods measured using Wrist-wearable actigraphy | Baseline, 3 months and 6 months
  The amount of time spent sleep walking in naturalistic settings will be measured using the ActiGraph which will be worn on the non-dominant wrist for 24-hours each day for seven consecutive days.
Change in 24 hour ambulatory average systolic blood pressure | Baseline, 3 months and 6 months
  24-hour ambulatory blood pressure monitoring using a blood pressure monitoring device to measure average systolic blood pressure
Change in 24 hour ambulatory average diastolic blood pressure | Baseline, 3 months and 6 months
  24-hour ambulatory blood pressure monitoring using a blood pressure monitoring device to measure average diastolic blood pressure
Change in 24 hour ambulatory blood pressure variability | Baseline, 3 months and 6 months
  24-hour ambulatory blood pressure monitoring using a blood pressure monitoring device measure blood pressure variability over 24 hour monitoring session.
Change in 24 hour ambulatory nighttime blood pressure dipping | Baseline, 3 months and 6 months
  Comparing average BP during wakefulness to average BP during major sleep episode in 24 hours monitoring session
Change in Vdrive/Loop gain by aPSG | Baseline and 6 months
  Mathematical modeling to determine the patient's ventilatory drive (or desired ventilation, Vdrive) in response to changes in ventilation induced by upper airway obstruction (i.e., apnea/hypopnea). The Vdrive signal is fit to the ventilation (VE) signals when the airway is expected to be patent (VE = Vdrive). Recorded during the sleep study. Measures of Vdrive allow determinations of Loop gain (LG), measured by the increase in ventilatory drive that occurs following a unit reduction in ventilation due to apneas/hypopneas.
Vdrive/Arousal threshold (ArTH) by aPSG | Baseline and 6 months
  Mathematical modeling to determine the patient's ventilatory drive (or desired ventilation, Vdrive) in response to changes in ventilation induced by upper airway obstruction (i.e., apnea/hypopnea). The Vdrive signal is fit to the ventilation (VE) signals when the airway is expected to be patent (VE = Vdrive). Recorded during the sleep study. Measures of Vdrive allow determinations of Arousal threshold (ArTH), quantified as the level of "ventilatory drive" just before arousal from sleep.
Vdrive/Pharyngeal muscle compensation (Mresp) by aPSG | Baseline and 6 months
  Mathematical modeling to determine the patient's ventilatory drive (or desired ventilation, Vdrive) in response to changes in ventilation induced by upper airway obstruction (i.e., apnea/hypopnea). The Vdrive signal is fit to the ventilation (VE) signals when the airway is expected to be patent (VE = Vdrive). Recorded during the sleep study. Measures of Vdrive allow determinations of Pharyngeal muscle compensation (Mresp), assessed by the increase in ventilation achieved during sleep per unit increase in the ventilatory drive. The analysis is automated using custom MATLAB software.

CONTACTS AND LOCATIONS:
Overall Officials: Henry K Yaggi, M.D., Principal Investigator — Yale University; Ian J Neeland, M.D., Principal Investigator — Case Western Reserve University School of Medicine
Locations (2):
- United States (2):
  - Yale New Haven Health, New Haven, Connecticut
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No